CLINICAL TRIAL: NCT03445481
Title: Pilot Study of New Prosthesis for Trans-femoral Amputated Patients Clinical Study Protocol
Brief Title: Clinical Pilot Study of New Prosthesis for Trans-femoral Amputated Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Christian Candrian (Other)
Responsible Party: Sponsor-Investigator, Christian Candrian, MD, Ente Ospedaliero Cantonale, Bellinzona
Organization: Ente Ospedaliero Cantonale, Bellinzona (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ORL ORT 001
Record Dates: First submitted 2018-01-09; First posted 2018-02-26 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Trans-femoral Amputated Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Femoral prosthesis (Experimental): newly developed prosthesis for trans-femoral amputation
  Interventions: Device: Medacta femoral prosthesis

INTERVENTIONS:
Device: Medacta femoral prosthesis — patients' treatment with a new implant prosthesis

SUMMARY:
Patients with a trans-femoral amputation who experienced problems, complications pain due to the ischial weight bearing and discomfort with conventional socket prosthesis will be proposed to implant a new developed prosthesis.

DETAILED DESCRIPTION:
The patients will undergo a surgical operation to implant a femoral prosthesis according to the hospital's protocol. The surgical intervention will be performed under general or spinal anesthesia with a tourniquet at the root of the lower limb. Under sterile conditions, the incision of the stump will be done at the level of the previous surgical scar. Preserving the soft tissue, the distal femoral bone is reached. Then, the medullary canal is opened and prepared with reamers of increasing diameter. A femoral cemented stem of appropriate dimensions correlated to the size of the canal and 105 mm of height is implanted. To the above-mentioned stem, the Medacta prosthesis will be fixed with a blocking screw. The prosthesis is then covered with the soft tissue and layered suturing of the stump is performed.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 and <75 years
* Patients with Trans-femoral Amputations since at least 2 years and suffering from pain and discomfort with the current standard socket prosthesis, i.e., with a baseline VAS score for pain between 3 and 10 or a health-related quality of life (Eq-5D) score < 60 or an SF-36 result below the 50th percentile
* Amputation due to:

  1. Trauma
  2. Oncologic disease
* Written informed consent

Exclusion Criteria:

* Trans-femoral amputation due to infection
* Patients affected by

  1. metabolic disease
  2. neurologic degenerative disease
  3. vascular disease proximal to the amputation
  4. body weight >100 kg
  5. Hip arthritis of the amputated limb

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2018-02-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Quality of Life | Two years
  Patients outcome evaluation of health-related quality of life through quality of life questionnaire EQ-5D-5L

SECONDARY OUTCOMES:
Adverse Events | Two years
  Post surgery adverse events collecting adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Christian Candrian, Dr. med, Principal Investigator — EOC
Locations (1):
- Ospedale Regionale di Lugano Civico e Italiano, Lugano, Switzerland

IPD SHARING:
Plan to Share IPD: No
not foreseen